CLINICAL TRIAL: NCT01670994
Title: A Study of ALT-801 in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: QUILT-3.020: A Study of ALT-801 in Patients With Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Patient population did not benefit from single agent treatment.
Sponsor: Altor BioScience (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA-ALT-801-01-11
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Results first posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-05

CONDITIONS: Relapsed or Refractory Multiple Myeloma
Keywords: cancer; immunotherapy; immunochemotherapy; targeted; metastatic; interleukin-2; antitumor; TCR; T-cell receptor; p53; p53 gene; p53 tumor supressor protein; HLA-A2 positive; HLA-A*0201/p53 aa264-272; HLA complex; multiple myeloma; IFN-γ and TNF-α; refractory; relapsed
MeSH Terms: conditions — Recurrence; Multiple Myeloma; Neoplasms; Neoplasm Metastasis | interventions — ALT-801

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALT-801 0.04mg/kg (Experimental)
  Interventions: Biological: ALT-801
- ALT-801 0.06mg/kg (Experimental)
  Interventions: Biological: ALT-801

INTERVENTIONS:
Biological: ALT-801 — Intravenous infusion; 2 treatment cycles: on day 1, 3, 8, and 15 of each cycle
  Other Names: c264scTCR-IL2

SUMMARY:
This is a Phase Ib/II, open-label, multi-center and competitive enrollment study of ALT-801 in patients who have relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
Multiple Myeloma (MM) is a plasma cell malignancy that makes up 1% of all cancers and 10% of hematologic neoplasma, and is the second most commonly diagnosed hematologic malignancy. There are an estimated 20,520 new cases of MM and 10,610 deaths due to MM in the United States. Historically, standard first-line therapy for MM consisted of combination therapy with an alkylating agent, such as melphalan and prednisone. Response rates with such combination therapy are approximately 50%, but five-year survival rates remain low at 33%. For younger patients, debulking chemotherapy followed by autologous stem cell transplant (ASCT) with melphalan is the treatment of choice to increase the potential for a sustained durable remission. However, a large percentage of patients diagnosed with MM are not suitable candidates for ASCT because of age or comorbidities. The approach to MM treatment has undergone a radical transformation over the past decade with the introduction of the proteasome inhibitor, bortezomib, and immunomodulatory drugs (ImiDs), thalidomide or lenalidomide. Despite some advances in the treatment of MM, the disease remains incurable due to the persistence of minimal residual disease. Thus, novel modalities complementing or improving current treatment options are needed.

There is ample evidence that immunomodulatory drugs are effective against myeloma. Lenalidomide and thalidomide have been shown to stimulate T cells in the presence of antigen presenting cells via costimulatory pathway. Also, modulation of NK cell function has been associated with anti-tumor activity observed in MM patients treated with lenalidomide. It has been demonstrated that NK cells exhibit potent anti-MM activity following IL-2 administration, and ex vivo IL-2-activated and intravenously administered NK cells prolong survival in MM-bearing mice. Thus further demonstrating the role and importance of NK cells in the treatment of MM. Taken together, these data suggest that the use of a potent immunotherapeutic is an attractive approach to provide durable immune responses to or even potentially curing patients with MM.

Additionally, immunotherapy is a well-established approach for treating other cancer types. One strategy that has received attention is treatment with cytokines such as IL-2 to enhance anti-tumor immunity. Unfortunately, the considerable toxicity associated with this treatment makes it difficult to achieve an effective dose at the site of the tumor and limits the population that can be treated. Thus, there is a critical need for innovative strategies that enhance the effects of IL-2, reduce its toxicity without compromising clinical benefit, provide a more convenient dosing regimen, and treat other diagnoses including MM.

Altor Bioscience Corp. has developed a tumor-targeted IL-2 fusion protein, ALT-801, comprising human recombinant IL-2 genetically linked to a TCR domain capable of binding a tumor associated human p53 peptide presented in the context of HLA-A2.

ELIGIBILITY:
ENTRY CRITERIA:

DISEASE CHARATERISTICS:

* Confirmed diagnosis of relapsed/refractory multiple myeloma after treatment with at least two different previous regimens.

  * Refractory disease is defined as progressive disease while on therapy or progression within 60 days of therapy.
  * Progressive disease is defined by a 25% increase from the lowest response value in specified tests.
* Measurable disease as defined by at least one of the following:

  * Serum M-protein ≥ 1g/dL (for IgG, IgM) or 0.5 g/dL (for IgA)
  * Urine M-protein ≥ 200mg/24hours
  * Serum free light chains ≥ 10 mg/dL and abnormal kappa/lambda ratio

PRIOR/CONCURRENT THERAPY:

* No anti-myeloma treatments within 28 days before the start of study treatment.
* Must have recovered from side effects of prior treatments.

PATIENT CHARACTERISTICS:

Age

• ≥ 18 years

Performance Status

• ECOG 0, 1, or 2

Bone Marrow Reserve

* Absolute neutrophil count (AGC/ANC) ≥ 1,000/uL
* Platelets ≥ 30,000/uL
* Hemoglobin ≥ 8g/dL

Renal Function

• Glomerular Filtration Rate (GFR) > 45mL/min/1.73m^2

Hepatic Function

* Total bilirubin ≤ 2.0 X ULN
* AST, ALT, ALP ≤ 3.0 X ULN, or ≤ 5.0 X ULN (if liver metastases exist)

Cardiovascular

* No congestive heart failure < 6 months
* No unstable angina pectoris < 6 months
* No myocardial infarction < 6 months
* No history of ventricular arrhythmias
* No history of supraventricular arrhythmias
* No NYHA Class > II CHF
* Normal Transthoracic Echocardiogram (TTE) is required for patients with history of EKG abnormalities, CHF, coronary artery disease or other cardiac disease, or with a history of having received adriamycin or doxorubicin
* Patients with a left ventricular ejection fraction (LVEF) of less than 50% will be excluded from study entry

Pulmonary

• Normal clinical assessment of pulmonary function

Other

* Negative serum pregnancy test if female and of childbearing potential
* Women who are not pregnant or nursing
* Subjects, both females and males, with reproductive potential must agree to use effective contraceptive measures for the duration of the study
* No known autoimmune disease other than corrected hypothyroidism
* No known prior organ allograft or allogeneic transplantation
* Not HIV positive
* No history or evidence of uncontrollable CNS disease
* No psychiatric illness/social situation
* No other illness that in the opinion of the investigator would exclude the subject from participating in the study
* Must provide informed consent and HIPPA authorization and agree to comply with all protocol-specified procedures and follow-up evaluations
* Active systemic infection requiring parenteral antibiotic therapy.
* No ongoing chronic systemic steroid therapy required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-08-14 (Actual); Primary Completion 2015-09-09 (Actual); Study Completion 2015-09-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Hospitals, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only the Phase 1b portion of the study enrolled participants. The study was terminated early, so no participants were enrolled on the Phase 2 portion of the study.
Period: Overall Study
Arm/Group | ALT-801 0.04mg/kg | ALT-801 0.06mg/kg
Started | 3 | 3
Completed | 3 | 0
Not Completed | 0 | 3
Not completed — Disease Progression and Switched to Alternative Treatment | 0 | 1
Not completed — Disease Progression and Did Not Qualify or Consent for Repeat Treatment | 0 | 1
Not completed — Patient experienced DLT | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ALT-801 0.04mg/kg | ALT-801 0.06mg/kg | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (6.9) | 64 (4.0) | 66 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Patients with Relapsed or Refractory Multiple Myeloma [Count of Participants; unit: Participants] | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Related Adverse Events
Description: Number of treatment related AEs that occur or worsen after the first dose of study treatment
Time Frame: 7 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ALT-801 0.04mg/kg | ALT-801 0.06mg/kg
Number analyzed (Participants) | 3 | 3
Participants | 3 | 3

ADVERSE EVENTS:
Time Frame: From start of treatment up to 72 days
Arm/Group | ALT-801 0.04mg/kg | ALT-801 0.06mg/kg
All-Cause Mortality (participants affected / at risk) | 1/3 | 3/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALT-801 0.04mg/kg (N=3) | ALT-801 0.06mg/kg (N=3)
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ALT-801 0.04mg/kg (N=3) | ALT-801 0.06mg/kg (N=3)
Influenza like illness (General disorders) | 3 | 2
Oedema peripheral (General disorders) | 3 | 1
Fatigue (General disorders) | 1 | 2
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Platelet count decreased (Investigations) | 2 | 2
Neutrophil count decreased (Investigations) | 1 | 1
Weight decreased (Investigations) | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Akathisia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Irritability (Psychiatric disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 1
Flushing (Vascular disorders) | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Cataract (Eye disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-01-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT01670994/Prot_SAP_000.pdf